CLINICAL TRIAL: NCT07086183
Title: Assessing Surgical Perioperative rIsk in Patients on chRonic aspIrN Therapy Undergoing Elective Craniotomy for Aneurysm Clipping: a Prospective Multi-center Observational Study (ASPIRIN)
Brief Title: Perioperative Risk in Patients on Chronic Aspirin Undergoing Craniotomy
Acronym: ASPRIN
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shaun Gruenbaum, Principal Investigator, Mayo Clinic
Other Study IDs: 25-006605
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Aneurysm Cerebral
Keywords: craniotomy; aneurysm clipping; aspirin; postoperative bleeding
MeSH Terms: conditions — Intracranial Aneurysm; Postoperative Hemorrhage | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic aspirin: Patients on chronic aspirin
  Interventions: Other: Observation
- No aspirin: Patients who are not on aspirin
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of intraoperative and postoperative outcomes

SUMMARY:
This study is looking at how taking aspirin regularly affects bleeding during and after brain surgery. Specifically, it focuses on patients who are having elective surgery to clip a brain aneurysm.

Aspirin is commonly used to prevent heart attacks and strokes, but it can also increase the risk of bleeding. Doctors often face a tough decision: should patients stop taking aspirin before surgery to reduce bleeding risk, or continue it to prevent blood clots?

To help answer this question, researchers will observe 100 patients, some who take aspirin regularly and some who don't, at hospitals in the U.S., Russia, and Italy. They will not change any treatments but will collect information about bleeding during surgery, blood test results, and CT scans after surgery.

The goal is to better understand the risks of continuing aspirin and to help doctors make safer decisions for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Patients willing to participate and provide an informed consent
* Patients undergoing elective craniotomy for cerebral aneurysm clipping
* Patients on chronic low-dose (75-100 mg) aspirin daily (aspirin group) or not on aspirin therapy for at least 7 days (control group) preoperatively.

Exclusion Criteria:

* Emergency craniotomy
* Use of other antiplatelet or anticoagulant medications within 7 days prior to surgery
* Known bleeding disorders (e.g. hemophilia, thrombocytopenia)
* History of intracranial hemorrhage unrelated to aneurysm
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective craniotomy for cerebral aneurysm clipping
  Recruited from three international sites:
  Mayo Clinic Florida (USA) Burdenko National Medical Research Center of Neurosurgery (Russia) Sapienza University of Rome (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Hemorrhage Rate | 48 hours postoperatively
  The incidence of postoperative hemorrhage detected on CT scans within 48 hours after surgery.
Intraoperative Blood Loss | From start to end of surgery
  Measured by the change in hemoglobin and hematocrit levels from preoperative baseline to immediate postoperative period.

SECONDARY OUTCOMES:
Subjective Bleeding Severity | From start to end of surgery
  Rated by the operating surgeon using a standardized 5-point Likert scale (0 = no bleeding to 4 = severe bleeding)
Need for Blood Transfusion | From start of surgery to day of discharge, up to 7 days
  The number of patients requiring intraoperative or postoperative blood transfusions.
Length of hospital stay | From end of surgery to day of discharge, up to 7 days
  Duration of hospitalization from the day of surgery to discharge
Surgical complications | From end of surgery to day of discharge, up to 7 days
  Incidence of surgical complications such as infection or reoperation.

CONTACTS AND LOCATIONS:
Locations (3):
- Mayo Clinic Florida, Jacksonville, Florida, United States
- Sapienza University of Rome, Roma, Italy
- Burdenko National Medical Research Center of Neurosurgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No